CLINICAL TRIAL: NCT03607032
Title: Evaluation of the Efficacy and Safety of the Use of the RespIn PAD in the Bronchial De-enclosure of Elderly Patients Who Cannot Benefit From Respiratory Physiotherapy
Brief Title: Use of RespinPAD in Elderly Patients
Acronym: RESPINPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-PP-17
Record Dates: First submitted 2018-02-15; First posted 2018-07-31 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Acute or Chronic Respiratory Pathologies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RespinPad and usual treatment (Experimental)
  Interventions: Device: Respin Pad; Other: usual treatment
- only usual treatment (Active Comparator)
  Interventions: Other: usual treatment

INTERVENTIONS:
Device: Respin Pad — RespinPad slid into the back of the patient sitting at 45° in the armchair or bed.
  Arms: RespinPad and usual treatment
Other: usual treatment — medical aerosol session followed by aspiration or not, as required

SUMMARY:
Secretive (or obstructive), acute or chronic pathologies are common in an increasing number of elderly patients. The medical teams are confronted with difficulties in the management of these patients: they do not benefit from optimal respiratory physiotherapy, whether manual or mechanical, due to functional deficiencies, cognitive functions that are sometimes limited or poorly adapted equipment.

The objective of this pilot study is to evaluate the effectiveness of a new RespinPAD device in the bronchial de-encapsulation of elderly patients who cannot benefit from optimal physiotherapy compared to conventional treatment (nasal or bucco-tracheal aspiration and aerosols).

The study will include 20 non-dementia patients and 20 dementia patients who will benefit from the use of RespinPAD and 20 patients who will benefit from conventional therapy. All the patients included will be over 70 years old and will be recruited when they are admitted to hospital in the geriatric hospital of the CHU de Nice. They will be included if they present a bronchial obstruction secondary to a respiratory pathology secreting whatever the etiology and for which optimal respiratory physiotherapy is not possible after evaluation by a physiotherapist.

Patients using the RespinPAD device will benefit from a 20-minute session twice daily for 5 days.

The primary endpoint (quantitative criterion) will be the measurement of oxygen consumption (VO2) and carbon dioxide production (VCO2) volumes for each patient included before and after each session of RespinPAD use or conventional treatment for the control group.

Secondary judging criteria will be a heteroassessment of the SEVA (Airway Overcrowding Score), the Borg Scale and the Algoplus or Digital Comfort Scale. For the effectiveness assessment, the SEVA score will allow for a qualitative assessment to complement the primary endpoint. The collection of volumes of secretions, pulse oximeter, mean length of stay, O2 withdrawal time and drug aerosols will also be used to compare results with previous studies. With regard to secondary safety and feasibility criteria, hemodynamic constants, electrocardiogram and the actual duration of the sessions will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 70 years of age
* member of the social security system
* hospitalized at the gerontology centre of the CHU de Nice (Cimiez): short geriatric stay, follow-up care and rehabilitation, long-term care unit or EHPAD.
* presenting a clinical bronchial obstruction (auscultatory signs with ronchi type) secondary to a secreting pathology (exacerbation of asthma or chronic obstructive bronchitis, acute bronchitis or acute infectious pneumonitis, repeated swallowing disorders, pulmonary disease of inhalation...) with or without radiological bronchial syndrome.
* for which a respiratory physiotherapy is not effective after expertise of the physiotherapist

Exclusion Criteria:

* a patient who is not hemodynamically stable or who has impaired alertness (glasgow<15) or shows signs of respiratory control (choracic-abdominal sway, costal or superclavicular draft, bronchospasm),
* Patient or trustworthy person who did not complete and sign the consent to participate in the study,
* a patient with chest pain, clinical intracranial hypertension (HIC) greater than 20 mmHg, uncontrolled high blood pressure, dyspnea of a different etiology than bronchial obstruction (a rapid and/or poorly tolerated ACFA, clinical or radiological pleural effusion, empyema, pneumothorax, decompensated heart failure, pericarditis, pericarditis
* The patient cannot benefit from naso-tracheal aspiration,
* End-stage palliative care patient
* patient already participating in another study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2020-10-24 (Actual)

PRIMARY OUTCOMES:
VO2 | 17 months
  Measurements of oxygen consumption (VO2) (quantitative) volumes on each patient included before and after each RespinPad session, and before and after each conventional treatment for the control group.
VCO2 | 17 months
  Measurements of carbon dioxide production (VCO2) (quantitative) volumes on each patient included before and after each RespinPad session, and before and after each conventional treatment for the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No